CLINICAL TRIAL: NCT02060734
Title: Lidocaine Injection Versus Sham Needling in Treating Whiplash Associated disorder-a Randomized Controlled Trial
Brief Title: Lidocaine Injection Versus Sham Needling in Treating Whiplash Associated Disorder
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: no participant recruited
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Maggie Qiyun Shi, Graduate student, Western University, Hamilton Health Sciences Corporation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HHSCTRIGGERINJ1402
Record Dates: First submitted 2014-02-07; First posted 2014-02-12 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2015-08

CONDITIONS: Whiplash Injuries; Neck Pain
Keywords: Whiplash,; injection,; lidocaine,; sham needling
MeSH Terms: conditions — Whiplash Injuries; Neck Pain | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- lidocaine (Experimental): The treatment group will receive a 25 gauge, 40mm long needle, pre-filled with 1% lidocaine inserting into the site of the trigger point. Three to five points injection.
  Interventions: Procedure: Lidocaine
- Saline (Active Comparator): The control group will receive a 25 gauge, 40mm long needle, pre-filled with saline inserting to subcutis.
  Interventions: Other: Saline

INTERVENTIONS:
Procedure: Lidocaine — Lidocaine injection 3-5 points in experimental group( using 25 gauge, 40mm long needle, pre-filled with 1% lidocaine inserting into the site of the trigger point).
  Arms: lidocaine
Other: Saline — The control group will receive a 25 gauge, 40mm long needle, pre-filled with saline inserting to subcutis.
  Arms: Saline

SUMMARY:
To determine the efficacy of lidocaine injection of trigger points versus subcutaneous injection in patients with subacute whiplash associated disorder following injury.

DETAILED DESCRIPTION:
This is a double-blind, randomized controlled trial to determine the efficacy of lidocaine injection of trigger points versus subcutaneous injection in patients with subacute whiplash associated disorder following injury. Outcomes include pain, objective assessment, self-report function recovery, impact on work performance and globe perceived effects which will be assessed 5 minutes, 2 and 6 weeks following injection.

ELIGIBILITY:
Inclusion Criteria:

* fulfill the Grade II Quebec Task Force classification of WAD,
* with identifiable myofascial trigger points ( which occur with or without a taut band),
* reproduction of recognizable pain with sustained pressure ( up to 10 seconds) on trigger points
* aged 18 to 70
* a good understanding of informed consent and willing to attend this trial.

Exclusion Criteria:

* have serious injury such as fracture and internal bleeding
* suspicion of upper cervical instability or neurological deficits
* clinical evidence of radiculopathy
* a history of active cancer, central nerve disorder, blood clotting disorders, needle phobia
* anticoagulant medication user
* previous experience with any type of needling for myofascial pain

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2016-01 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
pain | 2 weeks following injection
  10 cm Visual Analog Scale

SECONDARY OUTCOMES:
cervical range of motion | Immediately, 2 and 6 weeks after injection
self-report neck disability | Immediately, 2 and 6 weeks after injection
globe perceived effects | Immediately, 2 and 6 weeks after injection
  The Short Form-12
work performance | Immediately, 2 and 6 weeks after injection
  questionnaire
pain | 5 minutes following injection
  10 cm Visual Analog Scale
pain | 6 weeks following injection
  10 cm Visual Analog Scale

CONTACTS AND LOCATIONS:
Overall Officials: Joy MacDermid, Ph.D., Study Director — McMaster University
Locations (2):
- Canada (2):
  - Department of physical medicine and rehabilitation, McMaster University, Hamilton, Ontario
  - HHS (Juravinski Hospital Site), Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No